CLINICAL TRIAL: NCT04001101
Title: A Randomized Phase II Study of Anti-PD-1 and Limited Metastatic Site Radiation Therapy Versus Anti-PD-1 Alone for Patients With Microsatellite Instability-high (MSI-H) and Mismatch Repair Deficient (dMMR) Metastatic Solid Tumors
Brief Title: Anti-PD-1 +/- RT for MSI-H Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI has decided to withdraw the study
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0556.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-27 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Microsatellite Instability High; Mismatch Repair Deficiency; Colorectal Cancer
Keywords: Solid tumor; Colorectal cancer; Unresectable or metastatic
MeSH Terms: conditions — Turcot syndrome; Colorectal Neoplasms; Neoplasm Metastasis | interventions — spartalizumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In an effort to minimize bias, the study will utilize a randomization. The randomization list will be generated by the study biostatistician and provided only to the study personnel who will be responsible for assigning each subject to a cohort of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RT and Anti-PD-1 (Active Comparator): In the pembrolizumab + RT arm, pembrolizumab will be started on study within 7 days (+/- 7 days) of start of RT.
  Pembrolizumab will be given as standard of care in both arms
  Interventions: Combination Product: RT and Anti-PD-1
- Anti-PD-1 (Placebo Comparator): anti-PD-1 therapy alone Pembrolizumab will be given as standard of care in both arms
  Interventions: Drug: Anti-PD-1

INTERVENTIONS:
Combination Product: RT and Anti-PD-1 — limited metastatic site radiation
  Arms: RT and Anti-PD-1
Drug: Anti-PD-1 — anti-PD-1 therapy alone
  Arms: Anti-PD-1

SUMMARY:
To determine if the out-of-field ORR is improved with the addition of radiation therapy to anti-PD-1 for patients with MSI-H/dMMR metastatic solid tumors. Determine the rates of in-field tumor control, disease control (stable disease, partial response, complete response), durability of disease response, progression-free survival, overall survival, and to assess quality of life and toxicity. Determine the chronology and profile of the radiation-associated immune response.

DETAILED DESCRIPTION:
This is a randomized phase II study with a primary objective to compare the objective response rate (ORR) for anti-PD-1 therapy alone versus anti-PD-1 therapy and limited metastatic site radiation, in patients with microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) metastatic solid tumors. The anti-PD-1 agent, pembrolizumab, received recent FDA accelerated approval for the use in patients with metastatic MSI-H or dMMR solid tumors that have progressed following prior treatment or without satisfactory alternative treatment options. FDA approval for pembrolizumab was based on the results of five multi-cohort, multi-center, single-arm trials, which together showed an ORR of 39.6% among 149 patients with MSI-H/dMMR cancers. Importantly, there is mounting preclinical and clinic evidence supporting the safety and efficacy of combining radiation therapy with systemic immunotherapy, although no prospective comparative data, to the best of our knowledge. In this study, the investigators will focus on patients with MSI-H/dMMR tumors, given their baseline responsiveness to immune checkpoint inhibition, and test the hypothesis that ORR will be improved with radiation and anti-PD-1 therapy compared to anti-PD-1 therapy alone, through a randomized phase II trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Adult patients, 18-100 years of age.
4. ECOG 0 or 1.
5. Unresectable or metastatic MSI-H/dMMR tumors eligible to receive pembrolizumab according to FDA-approved indications:

   * Solid tumors that have progressed following prior treatment and who have no satisfactory alternative treatment options OR
   * Colorectal cancer that has progressed following treatment with a fluoropyrimidine, oxaliplatin, and irinotecan11
6. Confirmation from medical or gynecologic oncology that the patient is eligible to receive pembrolizumab per FDA-approved indication for patients not currently receiving pembrolizumab .
7. At least one site of disease amenable to radiation therapy per the acceptable dosing regimens outlined in section 6.2, and at least one additional site of measurable disease suitable for out-of-field response assessment.
8. Adequate baseline labs for initiation of trial treatment:

   * absolute neutrophil count (ANC) >1,000/µL
   * platelets >75,000/µL
   * hemoglobin >8 g/dL
   * serum creatinine < 1.5 x ULN
   * serum total bilirubin < 1.5 x ULN
   * AST and ALT < 2.5 x ULN, or < 5 x ULN if liver metastasis are present

Exclusion Criteria:

1. Pregnant women. Pregnancy testing is required for all female subjects of childbearing potential.
2. Patients with active collagen vascular disease (CVD), specifically systemic lupus erythematosus or scleroderma. Patients with a history of CVD without evidence of active disease are eligible for enrollment at the discretion of the study PI.
3. History of immunodeficiency, hypersensitivity to pembrolizumab, or other medical contraindication to receipt of pembrolizumab.
4. Active infection.
5. Active CNS metastases. Patients with treated CNS metastases are eligible.
6. Patients with a separate non-cutaneous cancer diagnosis for which the patient has not been without evidence of disease for at least 5 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Out-of-field ORR improvement | 12 months
  • Out-of-field objective response rate (ORR: CR+PR) according to RECIST 1.1 assessment

SECONDARY OUTCOMES:
in-field tumor control and disease control | 12 Months
  In-field tumor control and disease control will be defined as SD, PR, or CR, of the target lesion, by RECIST 1.1 criteria
Determine the chronology and profile of the radiation-associated immune response. | 12 months
  The University of Colorado School of Medicine Human Immune Monitoring Shared Resource (HIMSR) will quantify peripheral CD8, CD4, and regulatory T cell populations and characterize the relative functional state of these cells using activation markers (CD45RO, ICOS, and CD25) and inhibitory markers (TIM-3, CTLA-4, LAG-3, and PD-1). The HIMSR will also characterize peripheral dendritic cells (pDCs, CD1c+, and CD141+ subsets), monocytes (classical and non-classical subsets), myeloid-derived suppressor cells (MDSCs, granulocytic and monocytic subsets), and expression of activation (CD80 and HLA-DR) and inhibitory molecules (PDL1) on these cells. Further, cytokine production by NK cells, B cells, T cells, and monocytes will be measured by flow cytometry after brief ex-vivo stimulation. The HIMSR will also perform a protein multiplex array of 40 potential biomarkers in plasma.
Durability of disease response | 12 months
  In patients that achieve an objective response to pembrolizumab +/- RT, durability of response will be measured from the initiation of pembrolizumab until PD.
Progression-free Survival | 12 months
  Progression-free survival will be measured from the date of initiation of pembrolizumab to the time of tumor progression or death from any cause for one year.
Overall Survival | 12 Months
  Overall survival will be measured from the date of initiation of pembrolizumab to the time of death from any cause for one year.
Quality of life score | 12 Months
  Quality of life questionnaire, 28 questions rating experience from 1 to 4 (4 being "very much", 1 being "not at all") and two questions rating overall health and quality of life on a scale from 1 to 7 (7 being excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No